CLINICAL TRIAL: NCT03860181
Title: Investigation of a New Skin Closure Device, Dermabond PRINEO, for Total Shoulder Arthroplasty: A Randomized, Controlled Trial
Brief Title: Dermabond PRINEO for Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Josef Eichinger, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00084714
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Surgical Wound; Shoulder Arthritis; Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Traditional Dermabond + subcuticular sutures - Surgeon 1 (Active Comparator): Subcuticular sutures with traditional Dermabond applied to incision.
  Interventions: Procedure: Subcuticular Sutures - Surgeon 1
- Metal staples - Surgeon 2 (Active Comparator): Metal staples
  Interventions: Procedure: Metal Staples - Surgeon 2
- Dermabond PRINEO - Surgeon 1 (Experimental): Dermabond PRINEO System
  Interventions: Device: PRINEO - Surgeon 1
- Dermabond PRINEO - Surgeon 2 (Experimental): Dermabond PRINEO System
  Interventions: Device: PRINEO - Surgeon 2

INTERVENTIONS:
Procedure: Subcuticular Sutures - Surgeon 1 — This intervention closes incisions after shoulder arthroplasty using subcuticular sutures with Dermabond.The deep layer closure will require interrupted sutures.
  Arms: Traditional Dermabond + subcuticular sutures - Surgeon 1
Procedure: Metal Staples - Surgeon 2 — This intervention closes incisions after shoulder arthroplasty with metal staples. The deep layer closure will require interrupted sutures,
  Arms: Metal staples - Surgeon 2
Device: PRINEO - Surgeon 1 — The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
  Arms: Dermabond PRINEO - Surgeon 1
Device: PRINEO - Surgeon 2 — The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
  Arms: Dermabond PRINEO - Surgeon 2

SUMMARY:
This is a research study to find out whether wound closure (the process of closing the surgical wound after the procedure is complete) with Dermabond PRINEO Skin Closure System (PRINEO) will be faster and improve wound healing compared to standard closing methods after total shoulder replacement. The PRINEO system involves using running stitches to close the wound, and then taping over the sutures with a sticky film that holds the wound closed.

ELIGIBILITY:
Subjects will be included if:

* They are 18 years or older;
* They are undergoing primary total shoulder arthroplasty by the principal and co-investigator.
* They are willing and have the capacity to provide informed consent;
* They expect to continue their post-operative follow up care with their operating surgeons at Medical University of South Carolina (MUSC).

Subjects will be excluded if:

* They have a unique, identifying tattoo or skin marking within 2 inches of intended site of surgical incision
* They self-report a known hypersensitivity to cyanoacrylate, formaldehyde, benzalkonium chloride, or pressure sensitive adhesive;
* They self-report or have a documented prior ipsilateral shoulder arthroplasty or other open ipsilateral shoulder surgery utilizing the delto-pectoral approach;
* Their medical record shows that they are HIV positive or otherwise immunocompromised;
* Their medical record shows a skin abnormality or dermatological condition which affects skin healing;
* They report a personal or family history of significant keloid or significant hypertrophic scar formations, or other problems with wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Eichinger, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Dermabond + Subcuticular Sutures - Surgeon 1: Subcuticular sutures with traditional Dermabond applied to incision.
  Subcuticular Sutures: This intervention closes incisions after shoulder arthroplasty using subcuticular sutures with Dermabond.The deep layer closure will require interrupted sutures.
- Metal Staples - Surgeon 2: Metal staples
  Metal Staples: This intervention closes incisions after shoulder arthroplasty with metal staples. The deep layer closure will require interrupted sutures,
- Dermabond PRINEO - Surgeon 1; Dermabond PRINEO - Surgeon 2: Dermabond PRINEO System
  PRINEO: The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
Period: Overall Study
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Started | 21 | 22 | 25 | 21
Completed | 21 | 22 | 25 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2 | Total
Number analyzed (Participants) | 21 | 22 | 25 | 21 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 7 | 8 | 26
  >=65 years | 17 | 15 | 18 | 13 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 12 | 15 | 51
  Male | 8 | 11 | 13 | 6 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 1 | 1 | 6
  White | 21 | 18 | 24 | 20 | 83
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 25 | 21 | 89
Number of Participants Who Currently Smoke [Count of Participants; unit: Participants] — Patients who self-reported their smoking status as "Yes" at baseline.
  Participants | 0 | 2 | 4 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Total Cost of Wound Closure When Using Dermabond PRINEO Versus the Surgeon's Control.
Description: Closure cost was calculated by evaluating the cost of wound closure products ($) per patient, plus the cost of the operating room ($) per minute, multiplied by the closure time (minutes) per centimeter of incision length, then multiplied by the average incision length (cm) per patient.
Time Frame: 3 months post-operative
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 21 | 22 | 25 | 21
Dollars | 627.83 (90.22) | 304.75 (45.30) | 568.53 (88.98) | 420.77 (51.99)

2. Primary Outcome: Comparing Patient Satisfaction Ratings Between D.PRINEO and Controls
Description: Patient satisfaction ratings were on a scale from 0-10, where 0 = very dissatisfied and 10 = very satisfied.
Time Frame: 3 months post-operatively
Population: Participants who had adverse events before the conclusion of the study were excluded from this analysis, because outcome measures could not be collected.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 20 | 22 | 22 | 21
score on a scale | 10 [0 to 10] | 10 [0 to 10] | 10 [0 to 10] | 10 [0 to 10]

3. Primary Outcome: Mean Closure Time Per Centimeter of Incision
Description: This closure time was measured from the first stitch for closure to the application of the wound dressing. The incision length was measured immediately after closure.
Time Frame: Immediate/at time of surgery
Measure: Mean (Standard Error); unit: minutes/centimeters
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 21 | 22 | 25 | 21
minutes/centimeters | 1.3 (0.05) | 0.65 (0.02) | 1.1 (0.04) | 0.72 (0.03)

4. Secondary Outcome: Median Overall Opinion Score Reported by Operating Surgeon
Description: Overall Opinion was on a scale 1 - 10, where lower scores are viewed more favorably with 1=normal skin and 10=very different compared to adjacent skin, which was evaluated by the operating physician.
Time Frame: Up to 3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 20 | 22 | 22 | 21
score on a scale | 2 [1 to 10] | 1 [1 to 10] | 2 [1 to 10] | 1 [1 to 10]

5. Secondary Outcome: Median Wound Inflammation Score (AIRE) Reported by Operating Physician
Description: Images of the healing wound will be assessed according to the Acute Inflammatory Response Evaluation score (0 to 3, 0 being the lowest amount of inflammation and 3 represents the highest amount of inflammation) by the operating physician.
Time Frame: Up to 3 months post surgery
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 20 | 22 | 22 | 21
score on a scale | 0 [0 to 12] | 0 [0 to 12] | 0.5 [0 to 12] | 0 [0 to 12]

6. Secondary Outcome: Median Scar Assessment (POSAS) by Operating Surgeon
Description: Images of the healing wound will be assessed according to the Patient and Observer Scar Assessment Scale (POSAS, where there are six components each ranging between 1-10 with 10 representing the worst outcome, and each of those six components were summed for these results, having a final range of 6-60) by the operating surgeon.
Time Frame: Up to 3 months post surgery
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 20 | 22 | 22 | 21
score on a scale | 9 [6 to 60] | 6 [6 to 60] | 10 [6 to 60] | 6 [6 to 60]

7. Secondary Outcome: Wound Cosmesis (MHCS) Score by Operating Physician
Description: Evaluation of the wound after surgery will be assessed according to the Modified Hollander Cosmesis Scale (0 to 6, with 0 being ideal) by the operating physician.
Time Frame: Up to 3 months post surgery
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 20 | 22 | 22 | 21
score on a scale | 2 [0 to 6] | 1 [0 to 6] | 3 [0 to 6] | 1 [0 to 6]

8. Secondary Outcome: Differences Between Patient and Surgeon Total POSAS Scores
Description: POSAS scores can range from 1-10, where 1 is like normal skin, and 10 is worst scar imaginable, and has six components. Each component (range of 1-10) was summed up to get a final score (range of 6-60) for each participant. Differences were calculated as the participant's Patient and Observer Scar Assessment Scale (POSAS) score minus the physician POSAS score, with a negative difference signifying that the patients thought more highly of the scars than the physicians since lower POSAS scores are more favorable.
Time Frame: 3 months post-operatively
Population: Arms were regrouped to reflect the patient and surgeon scores for each intervention. Participants who had adverse events before the conclusion of the study were excluded from this analysis, because outcome measures could not be collected.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Traditional Dermabond + Subcuticular Sutures - Patient Scores: Patients that received the subcuticular sutures with traditional Dermabond applied for their incision intervention.
  Subcuticular Sutures: The intervention closes incisions after shoulder arthroplasty using subcuticular sutures with Dermabond. The deep layer closure will require interrupted sutures.
- Traditional Dermabond + Subcuticular Sutures - Surgeon 1 Scores: Surgeon 1 scores for patients who received Subcuticular sutures with traditional Dermabond applied to incision.
- Metal Staples - Patient Scores: Patients that received the metal staples intervention for their wound closure.
  Metal Staples: This intervention closes incisions after shoulder arthroplasty with metal staples. The deep layer closure will require interrupted sutures.
- Metal Staples - Surgeon 2 Scores: Surgeon 2 Scores for patients that received metal staples.
- Dermabond PRINEO - Surgeon 1 Patient Scores: Patients that received the Dermabond PRINEO System intervention for wound closure from Surgeon 1.
  PRINEO: The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
- Dermabond PRINEO - Surgeon 1 Scores: Surgeon 1 Scores for patients that received the Dermabond PRINEO closure system.
- Dermabond PRINEO - Surgeon 2 Patient Scores: Patients that received the Dermabond PRINEO System intervention wound closure from Surgeon 2.
  PRINEO: The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
- Dermabond PRINEO - Surgeon 2 Scores: Surgeon 2 Scores for patients that received the Dermabond PRINEO closure system.
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Patient Scores | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 Scores | Metal Staples - Patient Scores | Metal Staples - Surgeon 2 Scores | Dermabond PRINEO - Surgeon 1 Patient Scores | Dermabond PRINEO - Surgeon 1 Scores | Dermabond PRINEO - Surgeon 2 Patient Scores | Dermabond PRINEO - Surgeon 2 Scores
Number analyzed (Participants) | 20 | 20 | 22 | 22 | 22 | 22 | 21 | 21
units on a scale | 11.5 [6 to 60] | 9 [6 to 60] | 7 [6 to 60] | 6 [6 to 60] | 13 [6 to 60] | 10 [6 to 60] | 9 [6 to 60] | 6 [6 to 60]
Statistical Analysis 1: Comparison: Traditional Dermabond + Subcuticular Sutures - Patient Scores vs Traditional Dermabond + Subcuticular Sutures - Surgeon 1 Scores vs Dermabond PRINEO - Surgeon 1 Patient Scores vs Dermabond PRINEO - Surgeon 1 Scores; Test type: Equivalence — The statistical significance's p-value was set at 0.05. For Surgeon 1's differences, they were calculated as patient POSAS score - surgeon POSAS score, with a negative difference signifying that the patients thought more highly of the scars than the physicians since lower POSAS scores are more favorable; p = 0.896, Wilcoxon (Mann-Whitney); Mann-Whitney U = 215
Statistical Analysis 2: Comparison: Metal Staples - Patient Scores vs Metal Staples - Surgeon 2 Scores vs Dermabond PRINEO - Surgeon 2 Patient Scores vs Dermabond PRINEO - Surgeon 2 Scores; Test type: Equivalence — The statistical significance's p-value was set at 0.05. For Surgeon 2's differences, they were calculated as patient POSAS score - surgeon POSAS score, with a negative difference signifying that the patients thought more highly of the scars than the physicians since lower POSAS scores are more favorable; p = 0.612, Wilcoxon (Mann-Whitney); Mann-Whitney U = 210

9. Secondary Outcome: Median Overall Opinion Score Reported by Plastic Surgeons
Description: Overall Opinion was on a scale 1 - 10, where lower scores are viewed more favorably with 1=normal skin and 10=very different compared to adjacent skin, which was evaluated by an independent plastic surgeon.
Time Frame: Up to 3 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 19 | 22 | 21 | 20
score on a scale | 5 [1 to 10] | 3 [1 to 10] | 5 [1 to 10] | 4 [1 to 10]

10. Secondary Outcome: Median Scar Assessment (POSAS) by Plastic Surgeon
Description: Images of the healing wound will be assessed according to the Patient and Observer Scar Assessment Scale (POSAS, includes six measurements ranging from 0 to 10, 10 being ideal, where the total of the six measurements is what is reported) by an independent plastic surgeon. This POSAS total score would then range from 6-60.
Time Frame: Up to 3 months post surgery
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 19 | 22 | 21 | 20
score on a scale | 25 [6 to 60] | 18 [6 to 60] | 25 [6 to 60] | 20.5 [6 to 60]

11. Secondary Outcome: Wound Cosmesis (MHCS) Score by Plastic Surgeon
Description: Evaluation of the wound after surgery will be assessed according to the Modified Hollander Cosmesis Scale (0 to 6, with 0 being ideal) by an independent plastic surgeon.
Time Frame: Up to 3 months post surgery
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Traditional Dermabond + Subcuticular Sutures - Surgeon 1 | Metal Staples - Surgeon 2 | Dermabond PRINEO - Surgeon 1 | Dermabond PRINEO - Surgeon 2
Number analyzed (Participants) | 19 | 22 | 21 | 20
score on a scale | 2 [0 to 6] | 1 [0 to 6] | 3 [0 to 6] | 1 [0 to 6]

ADVERSE EVENTS:
Time Frame: The adverse even data was collected up to 3 months post-operatively.
Groups:
- Traditional Dermabond + Subcuticular Sutures: Subcuticular sutures with traditional Dermabond applied to incision.
  Subcuticular Sutures: This intervention closes incisions after shoulder arthroplasty using subcuticular sutures with Dermabond.The deep layer closure will require interrupted sutures.
- Metal Staples: Metal staples
  Metal Staples: This intervention closes incisions after shoulder arthroplasty with metal staples. The deep layer closure will require interrupted sutures,
- Dermabond PRINEO: Dermabond PRINEO System
  PRINEO: The closure system uses the Dermabond PRINEO (which is similar to clear tape stuck over the wound) placed over running sutures for both the deep and subcuticular layer.
Arm/Group | Traditional Dermabond + Subcuticular Sutures | Metal Staples | Dermabond PRINEO
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22 | 1/46
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Dermabond + Subcuticular Sutures (N=21) | Metal Staples (N=22) | Dermabond PRINEO (N=46)
Infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT03860181/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03860181/ICF_001.pdf